CLINICAL TRIAL: NCT04001374
Title: Platelet Sub-study of the TWILIGHT Trial
Status: Completed | Type: Observational
Sponsor: Juan Badimon (Other)
Responsible Party: Sponsor-Investigator, Juan Badimon, Professor of Medicine and Director of AtheroThrombosis Research Lab, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Other Study IDs: GCO 15-0769
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: Thrombosis; Platelets; Platelet Aggregation; Blood Thrombogenicity
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Thrombosis | interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ticagrelor: Ticagrelor 90mg tablet bid for 12 months
  Interventions: Drug: Ticagrelor
- Ticagrelor + ASA: Ticagrelor 90mg tablet bid for 12 months and enteric coated aspirin 81mg-100mg daily p.o. for 12 months
  Interventions: Drug: Ticagrelor; Drug: ASA

INTERVENTIONS:
Drug: Ticagrelor — 90mg tablet bid for 12 months
Drug: ASA — enteric coated aspirin 81mg-100mg daily p.o. for 12 months
  Groups: Ticagrelor + ASA

SUMMARY:
TWILIGHT study is a multicenter RCT comparing treatment with ticagrelor alone versus ticagrelor plus aspirin in high-risk patients after PCI. All patients will receive DAPT (ticagrelor plus aspirin) for the initial 3 months post-PCI and then be randomized to either Ticagrelor alone OR Ticagrelor plus Aspirin DAPT.

To investigate the pharmacodynamic effects of the two treatments in this trial, a 'Platelet Sub-study' will be conducted only at the Mount Sinai Medical Center. The sub-study will recruit randomized patients from the TWILIGHT Trial at Mount Sinai and conduct specialized blood tests at randomization and one month thereafter. The aim of the Platelet Sub-study is to compare the antithrombotic effects of Ticagrelor alone versus Ticagrelor plus Aspirin using an ex vivo model of thrombosis (Badimon Chamber).

DETAILED DESCRIPTION:
The present study will enroll a cohort of randomized patients from the TWILIGHT trial at the Mount Sinai Medical Center. These subjects will undergo blood sampling and measurement of thrombotic indices at the time of randomization and 1-6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in the TWILIGHT trial:

Clinical Inclusion Criteria (must meet at least one):

* Adult patients ≥ 65 years of age
* Troponin (+) acute coronary syndrome
* Female gender
* Established vascular disease defined as previous MI, documented PAD or CAD/PAD revascularization
* Diabetes mellitus treated with medications (oral hypoglycemic, subcutaneous injection of insulin)
* Chronic kidney disease defined as an estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73m2 or creatinine clearance (CrCl) < 60 ml/min

Angiographic Inclusion Criteria (must meet at least one):

* Multivessel coronary artery disease
* Target lesion requiring total stent length >30 mm
* Thrombotic target lesion(s)
* Bifurcation lesions with Medina X,1,1 classification requiring at least 2 stents
* Left main (≥50%) or proximal LAD (≥70%) lesion
* Calcified target lesion(s) requiring atherectomy

Exclusion Criteria:

Patients not eligible to participate in the TWILIGHT trial:

* Under 18 years of age
* Contraindication to aspirin
* Contraindication to ticagrelor
* Planned surgery within 90 days
* Planned coronary revascularization (surgical or percutaneous) within 90 days
* Need for chronic oral anticoagulation
* Prior stroke
* Dialysis-dependent renal failure
* Active bleeding or extreme-risk for major bleeding (e.g. active peptic ulcer disease, gastrointestinal pathology with a raised risk for bleeding, malignancies with a raised risk for bleeding)
* Emergent or salvage PCI or STEMI presentation.
* Liver cirrhosis
* Life expectancy < 1 year
* Unable or unwilling to provide informed consent
* Women of child bearing potential (as determined by hospital standard of care)
* Fibrinolytic therapy within 24 hours of index PCI
* Concomitant therapy with a strong cytochrome P-450 3A inhibitor or inducer
* Platelet count < 100,000 mm3
* Requiring ongoing treatment with aspirin > 325 mg daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Randomized subjects from the TWILIGHT trial treated at Mount Sinai Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-06-28 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Thrombus size (Badimon Chamber) | 1-6 months after randomization
  Thrombus area measured 1-6 months after randomization

SECONDARY OUTCOMES:
Platelet aggregation | 1-6 months after randomization
  Platelet aggregation assessed using Multiplate Analyzer 1-6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Juan Badimon, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baber U, Zafar MU, Dangas G, Escolar G, Angiolillo DJ, Sharma SK, Kini AS, Sartori S, Joyce L, Vogel B, Farhan S, Gurbel P, Gibson CM, Fuster V, Mehran R, Badimon JJ. Ticagrelor With or Without Aspirin After PCI: The TWILIGHT Platelet Substudy. J Am Coll Cardiol. 2020 Feb 18;75(6):578-586. doi: 10.1016/j.jacc.2019.11.056. PMID 32057371